CLINICAL TRIAL: NCT01579162
Title: Intra-Individual Reproducibility of the Non-Invasive Assessment of the Portal Circulation
Acronym: Repro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HepQuant, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HepQuant-001
Record Dates: First submitted 2012-02-09; First posted 2012-04-17 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Hepatitis C, Chronic; Non-Alcoholic Fatty Liver Disease
Keywords: Hepatitis; Fatty Liver
MeSH Terms: conditions — Hepatitis C, Chronic; Non-alcoholic Fatty Liver Disease; Hepatitis; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy Controls (Experimental): Healthy controls will be recruited to have approximately equal numbers of men and women. Controls will be of healthy weight as defined by a BMI 18-25 and without liver disease or risk factors for liver disease.
  Interventions: Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123)
- chronic HCV patients with F0-F2 fibrosis (Experimental)
  Interventions: Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123)
- chronic HCV patients with F3-F4 fibrosis (Experimental)
  Interventions: Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123)
- NASH patients with F0-F2 fibrosis (Experimental)
  Interventions: Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123)
- NASH patients with F3-F4 fibrosis (Experimental)
  Interventions: Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123)

INTERVENTIONS:
Device: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123) — The FDA has indicated that liver function diagnostic testing with stable isotope labeled cholates would be considered a drug/device combination product. The drugs administered at each test visit will be:
  20 mg Cholate-24-13C, IV (in the vein), dissolved in NaHCO3 and mixed with albumin.
  40 mg Cholate-2,2,4,4-d4, oral, dissolved in NaHCO3 and mixed with juice.
  The 3 test visits will be on separate days within a span of 30 days
  Other Names: Cholic acid-24-13C; Cholic acid-2,2,4,4-d4

SUMMARY:
HepQuant tests are new liver tests that are being developed to accurately measure liver function with sensitivity and specificity while being safe and non-invasive. The primary goal of this study is to define the intra-individual reproducibility of the HepQuant tests, that is, to see if a person is given the tests several times that the test results are essentially the same each time. Subjects for this study will include healthy controls and patients with chronic liver diseases. The chronic liver diseases will include hepatitis C virus (HCV) infection and a serious form of fatty liver disease, known as non-alcoholic steatohepatitis (NASH). The HCV and NASH patients will include men and women, and those with early stage and late stage liver disease as defined by the amount of fibrosis observed in their liver biopsies. Once a subject has been enrolled in the study they will be given the HepQuant tests on three separate days within the span of one month. The hypothesis of this study is that HepQuant tests will reproducibly report liver function in healthy controls and patients with all stages of chronic HCV and NASH liver disease and that liver function will decrease as the amount of liver fibrosis increases in the chronic liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic HCV or NASH
* Liver biopsy within 2 years of enrollment
* Compensated liver disease

Exclusion Criteria:

* Decompensated liver disease
* Currently being treated with beta blockers, ACE inhibitors, or other agents affecting FMD
* Malignancy diagnosed within 5 years of study enrollment without demonstrated clearance
* History of congestive heart failure
* Renal insufficiency with chronic kidney disease stage 4 or 5 (GFR < 30 mL/min/1.73m2)
* Crohn's disease or any active intestinal inflammatory condition
* Having an ileal resection
* Diabetic Gastroparesis
* Pregnancy or intent to become pregnant. Urine pregnancy tests will be performed at each visit.
* Inability to consent for one's self

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Burton, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Lauriski S, Curto TM, Stoddard A, Wright EC; HALT-C Trial Group. Quantitative liver function tests improve the prediction of clinical outcomes in chronic hepatitis C: results from the Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial. Hepatology. 2012 Apr;55(4):1019-29. doi: 10.1002/hep.24752. Epub 2012 Mar 1. PMID 22030902
- [Background] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Desanto JL, Curto TM, Wright EC; HALT-C Trial Group. Quantitative tests of liver function measure hepatic improvement after sustained virological response: results from the HALT-C trial. Aliment Pharmacol Ther. 2009 Mar 1;29(5):589-601. doi: 10.1111/j.1365-2036.2008.03908.x. Epub 2008 Dec 1. PMID 19053983
- [Background] Everson GT, Shiffman ML, Morgan TR, Hoefs JC, Sterling RK, Wagner DA, Kulig CC, Curto TM, Wright EC; Halt-C Trial Group. The spectrum of hepatic functional impairment in compensated chronic hepatitis C: results from the Hepatitis C Anti-viral Long-term Treatment against Cirrhosis Trial. Aliment Pharmacol Ther. 2008 May;27(9):798-809. doi: 10.1111/j.1365-2036.2008.03639.x. Epub 2008 Feb 7. PMID 18266997
- [Background] Everson GT, Martucci MA, Shiffman ML, Sterling RK, Morgan TR, Hoefs JC; HALT-C trial group. Portal-systemic shunting in patients with fibrosis or cirrhosis due to chronic hepatitis C: the minimal model for measuring cholate clearances and shunt. Aliment Pharmacol Ther. 2007 Aug 1;26(3):401-10. doi: 10.1111/j.1365-2036.2007.03389.x. PMID 17635375

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy controls will be recruited to have approximately equal numbers of men and women. Controls will be of healthy weight as defined by a BMI 18-25 and without liver disease or risk factors for liver disease.
  Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123): The FDA has indicated that liver function diagnostic testing with stable isotope labeled cholates would be considered a drug/device combination product. The drugs administered at each test visit will be:
  20 mg Cholate-24-13C, IV (in the vein), dissolved in NaHCO3 and mixed with albumin.
  40 mg Cholate-2,2,4,4-d4, oral, dissolved in NaHCO3 and mixed with juice.
  The 3 test visits will be on separate days within a span of 30 days
Period: Overall Study
Arm/Group | Healthy Controls | Chronic HCV Patients With F0-F2 Fibrosis | Chronic HCV Patients With F3-F4 Fibrosis | NASH Patients With F0-F2 Fibrosis | NASH Patients With F3-F4 Fibrosis
Started | 16 | 8 | 8 | 8 | 8
Completed | 16 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Chronic HCV Patients With F0-F2 Fibrosis | Chronic HCV Patients With F3-F4 Fibrosis | NASH Patients With F0-F2 Fibrosis | NASH Patients With F3-F4 Fibrosis | Total
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Full Range); unit: years] | 32.9 [24 to 62.7] | 54.9 [43 to 63] | 55.4 [44 to 62.4] | 45.9 [22 to 65] | 53.2 [47.7 to 59.6] | 48.4 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 2 | 5 | 4 | 20
  Male | 8 | 7 | 6 | 3 | 4 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 12 | 7 | 7 | 6 | 7 | 39
  Hispanic | 2 | 1 | 0 | 1 | 1 | 5
  Black | 1 | 0 | 1 | 0 | 0 | 2
  Unknown | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Cholate Shunt Test
Description: The Cholate Shunt Test result is defined as the ratio of the IV Cholate Clearance to the Oral Cholate Clearance and is expressed as a percentage. The higher the SHUNT percentage, the more the blood flow is shunting around the liver, the more severe the liver disease.
  The average of the SHUNT test results (ratio of IV Cholate Clearance to Oral Cholate Clearance) from all three time points (3 visits within 30 days) for each participant was used in the calculation of the group SHUNT Test results.
Time Frame: Average of all three study visits performed within 30 days
Measure: Mean (Standard Deviation); unit: SHUNT %
Groups:
- Chronic HCV Patients With F0-F4 Fibrosis; NASH Patients With F0-F4 Fibrosis: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123): The FDA has indicated that liver function diagnostic testing with stable isotope labeled cholates would be considered a drug/device combination product. The drugs administered at each test visit will be:
  20 mg Cholate-24-13C, IV (in the vein), dissolved in NaHCO3 and mixed with albumin.
  40 mg Cholate-2,2,4,4-d4, oral, dissolved in NaHCO3 and mixed with juice.
  The 3 test visits will be on separate days within a span of 30 days
Arm/Group | Healthy Controls | Chronic HCV Patients With F0-F4 Fibrosis | NASH Patients With F0-F4 Fibrosis
Number analyzed (Participants) | 16 | 16 | 16
SHUNT % | 28.0 (5.5) | 37.6 (11.6) | 33.4 (7.3)

2. Secondary Outcome: Intra-individual Reproducibility of the Cholate SHUNT Test Across All Subjects
Description: The intra-individual reproducibility of the Cholate Shunt Test (SHUNT %), will be defined by its average Coefficient of Variation (CV) and its Intra-Class Correlation (ICC). Each subject will be tested at baseline and then twice more on separate days within the span of one month. The CV of each subject's three replicate tests will be used to calculate the average CV for each type of test. All test results for each type of test will be used to calculate its ICC.
Time Frame: All three study visits within 30 days
Population: The goal of the analysis was to obtain the intra-individual results, so the subjects were not stratified by groups for this outcome measure.
Measure: Number (95% Confidence Interval); unit: ICC
Groups:
- All Subjects (Healthy, NASH, and Chronic HCV): All subjects recruited for this study - both Healthy and with HCV or NASH
  Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123): The FDA has indicated that liver function diagnostic testing with stable isotope labeled cholates would be considered a drug/device combination product. The drugs administered at each test visit will be:
  20 mg Cholate-24-13C, IV (in the vein), dissolved in NaHCO3 and mixed with albumin.
  40 mg Cholate-2,2,4,4-d4, oral, dissolved in NaHCO3 and mixed with juice.
  The 3 test visits will be on separate days within a span of 30 days
Arm/Group | All Subjects (Healthy, NASH, and Chronic HCV)
Number analyzed (Participants) | 48
ICC | 0.74 [0.63 to 0.84]

3. Secondary Outcome: Intra-class Reproducibility of the Disease Severity Index (DSI) by Histological Fibrosis Stage
Description: The intra-class correlation coefficients (ICCs) for reproducibility of the Disease Severity Index (DSI, an index value measuring severity of liver disease that can be calculated using the SHUNT Test results) were obtained by stage of liver fibrosis by liver biopsy.
  The DSI is a score on a scale from 0 (healthy) to 50 (severe liver disease), so the higher the DSI, the more severe the liver disease. Fibrosis scores increase with disease severity as well, so subjects with F0-F2 fibrosis have less severe liver disease than subjects with F3-F4 fibrosis.
Time Frame: Average of DSIs obtained from all three study visits within 30 days
Population: This analysis was conducted by histological fibrosis stage, so subjects with liver disease are grouped into two groups, either NASH & Chronic HCV patients with F0-F2 fibrosis or with F3-F4 fibrosis.
Measure: Number (95% Confidence Interval); unit: ICC
Groups:
- Nash + Chronic HCV Patients With F0-F2 Fibrosis; NASH + Chronic HCV Patients With F3-F4 Fibrosis: Cholate-24-13C (IND 65121) & Cholate-2,2,4,4-d4 (IND 65123): The FDA has indicated that liver function diagnostic testing with stable isotope labeled cholates would be considered a drug/device combination product. The drugs administered at each test visit will be:
  20 mg Cholate-24-13C, IV (in the vein), dissolved in NaHCO3 and mixed with albumin.
  40 mg Cholate-2,2,4,4-d4, oral, dissolved in NaHCO3 and mixed with juice.
  The 3 test visits will be on separate days within a span of 30 days
Arm/Group | Nash + Chronic HCV Patients With F0-F2 Fibrosis | NASH + Chronic HCV Patients With F3-F4 Fibrosis
Number analyzed (Participants) | 16 | 16
ICC | 0.840 [0.679 to 0.935] | 0.945 [0.880 to 0.979]

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | Healthy Controls | Chronic HCV Patients With F0-F2 Fibrosis | Chronic HCV Patients With F3-F4 Fibrosis | NASH Patients With F0-F2 Fibrosis | NASH Patients With F3-F4 Fibrosis
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes